CLINICAL TRIAL: NCT01945060
Title: Closed Loop Control in Adolescents Using Heart Rate as Exercise Indicator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Breton (Other)
Collaborators: Virginia Commonwealth University (Other); DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Marc Breton, Co-Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HM15215 & 17256; 17-2013-498 (Other Grant/Funding Number: JDRF)
Record Dates: First submitted 2013-09-10; First posted 2013-09-18 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas Project; Diabetes Assistant (DiAs) Medical Platform System; Artificial Pancreas Platform; Insulin Pump; Continuous Glucose Monitor; Closed-Loop Control; heart rate Control to Range System (hrCTR)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- heart rate Control to Range System (hrCTR) THEN No heart rate Control to Range System (hrCTR) (Experimental): The Diabetes Assistant (DiAs) Control-to-Range system is notified of heart rate during exercise. The study team member will activate and deactivate a heart rate button when the subject's heart rate exceeds and then returns below 140 beats per minute.
  Interventions: Device: heart rate Control to Range System (hrCTR) using DiAs Platform
- No heart rate Control to Range System (hrCTR) THEN heart rate Control to Range System (hrCTR) (Placebo Comparator): Using the DiAs Platform, the Control-to-Range system is not notified of the heart rate during exercise. Heart rate not of interest in this arm.
  Interventions: Device: heart rate Control to Range System (hrCTR) using DiAs Platform; Other: DiAs Control-to-Range System not informed for heart rate

INTERVENTIONS:
Device: heart rate Control to Range System (hrCTR) using DiAs Platform — Diabetes Assistant (DiAs) Medical Platform System
  * A smart-phone medical platform (DiAs);
  * Continuous Glucose Monitor;
  * Insulin pump;
  * Bluetooth connection;
  * Remote Monitoring Server.
Other: DiAs Control-to-Range System not informed for heart rate — Not informing system of heart rate during exercise.
  Arms: No heart rate Control to Range System (hrCTR) THEN heart rate Control to Range System (hrCTR)

SUMMARY:
The purpose of this study is to see if the Artificial Pancreas (AP) Platform can successfully control blood sugar in people with type 1 diabetes mellitus on insulin pump therapy in a hospital setting. Investigators will also be studying to see if the heart rate informed Control To Range (hrCTR) can improve the performance of the system during and immediately after exercise.

DETAILED DESCRIPTION:
The artificial pancreas (AP), known as Closed-Loop Control of blood glucose in diabetes, is a system combining a continuous glucose monitor (glucose sensor), a control algorithm (complex mathematical formulas), and an insulin pump. The algorithms are intended to maintain your blood glucose level within a certain range. This is called Control-to-Range. The algorithms are intended to maintain your blood glucose level within a certain range. The algorithms run on a portable AP platform on an Android smart phone, called the Diabetes Assistant (DiAs) Medical Platform.

In this study, researchers hypothesize that the heart rate informed Control To Range (hrCTR) will limit the risk for hypo and hyperglycemia during and immediately after exercise in adolescents 12 - 17 years of age and assess if the hrCTR will improve additional measures of overall short term glycemic control in this population.

This trial will be performed at both Virginia Commonwealth University and the University of Virginia. IRB approvals have been obtained at both institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for documented hyperglycemia (at least 1 must be met):

   * Fasting glucose ≥ 126 mg/dL - confirmed
   * Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥ 200 mg/dL - confirmed
   * Hemoglobin A1c (HbA1c) ≥ 6.5% documented - confirmed
   * Random glucose ≥ 200 mg/dL with symptoms
   * No data are available from the time of diagnosis but the participant has a convincing history of medical care and biochemical parameters consistent with T1DM
2. Criteria for requiring insulin at diagnosis (1 must be met):

   * Participant required insulin at diagnosis and continually thereafter
   * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did eventually require insulin that has been used continually
3. Criteria for Type 1 Diabetes Mellitus (T1DM) (at least 1 must be met):

   * Documented low or absent C-peptide level.
   * Documented presence of islet cell autoantibodies (ICA) or glutamic acid decarboxylase (GAD65) autoantibodies.
   * No data are available from the time of diagnosis but the participant has a convincing history of medical care and biochemical parameters consistent with T1DM

In addition, all subjects will meet the following additional criteria:

* Use an insulin pump (CSII) to treat his/her diabetes for at least 6 months
* Actively use a bolus calculator with the current insulin pump with pre-defined parameters for carbohydrate (CHO) ratio, insulin sensitivity factor (ISF), and target glucose
* Current HbA1c between 5.0% and 10.5% as measured with DCA2000 or equivalent device
* Not currently known to be pregnant, breast feeding, or intending to become pregnant (females)
* Demonstration of proper mental status and cognition for the study
* Willingness to avoid consumption of acetaminophen-containing products while wearing the continuous glucose monitor sensor.

Exclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes Mellitus (T2DM)
* Diabetic ketoacidosis within 6 months prior to enrollment
* Severe hypoglycemia resulting in seizure or loss of consciousness within 3 months prior to enrollment
* Pregnancy, breast feeding, or intention to become pregnant
* Subjects weighing less than 40 kg
* Hematocrit <36% (females); <38% (males)
* Conditions which may increase the risk of hypoglycemia such as known history of cerebrovascular event, history of arrhythmias, seizure disorder, syncope, adrenal insufficiency, or neurologic disease
* Additional conditions which may inhibit the ability to perform exercise (e.g. injury to or immobility of limbs, neuromuscular disease, exercise-induced asthma requiring inhaler use within the last 12 months or clinically impaired pulmonary function)
* Use of a medication that significantly lowers heart rate (beta blockers, reserpine, guanethidine, methyldopa, clonidine, cimetidine, digitalis, calcium channel blockers, amiodarone, antiarrythmic drugs, or lithium)
* History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the continuous glucose monitor (implantable cardioverter defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
* Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admission.
* Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment, uncontrolled anxiety or panic disorder)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Medical conditions that would make operating a continuous glucose monitor, cell phone or insulin pump difficult (e.g. blindness, severe arthritis, immobility)
* Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
* Known micro vascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment
* Active gastroparesis requiring current medical therapy
* If on antihypertensive, thyroid, or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Known bleeding diathesis or dyscrasia
* Allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor
* Anticoagulant therapy other than aspirin
* Oral steroids
* Active enrollment in another clinical trial
* Unwillingness to avoid acetaminophen while wearing the continuous glucose monitor sensor.
* Unwillingness to withhold dietary supplements two weeks prior to and during admission
* Unwillingness to use an approved form of birth control during this study by a sexually active female participant.
* Subject develops a febrile illness within 24 hours of inpatient admission.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Francis, MD, PhD, Principal Investigator — Virginia Commonwealth University; Marc Breton, PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

REFERENCES:
- [Result] DeBoer MD, Chernavvsky DR, Topchyan K, Kovatchev BP, Francis GL, Breton MD. Heart rate informed artificial pancreas system enhances glycemic control during exercise in adolescents with T1D. Pediatr Diabetes. 2017 Nov;18(7):540-546. doi: 10.1111/pedi.12454. Epub 2016 Oct 13. PMID 27734563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the University of Virginia and Virginia Commonwealth University from July 2013 through April 2015.
Pre-assignment Details: Of the 22 enrolled participants, 20 met inclusion criteria and were randomized to treatment. During the study, one participant withdrew from the trial because of distress related to intravenous access, and one participant did not finish the second admission within the allowed time window.
Groups:
- hrCTR THEN No hrCTR: The experimental admission (hrCTR) was defined as having the participant complete a exercise session where the Diabetes Assistant (DiAs) Control-to-Range system is notified of heart rate. The study team member activated and deactivated a heart rate button when the subject's heart rate exceeded and then returned below 140 beats per minute.
  The control admission (No hrCTR) had participants complete an exercise session where the closed loop is not informed about heart rate.
  Each admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
- No hrCTR THEN hrCTR: The control admission (No hrCTR) had participants complete an exercise session where the closed loop is not informed about heart rate.
  The experimental admission (hrCTR) was defined as having the participant complete a exercise session where the Diabetes Assistant (DiAs) Control-to-Range system is notified of heart rate. The study team member activated and deactivated a heart rate button when the subject's heart rate exceeded and then returned below 140 beats per minute.
  Each admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
Period: Overall Study
Arm/Group | hrCTR THEN No hrCTR | No hrCTR THEN hrCTR
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to follow up | 1 | 0
Not completed — Distress related to IV access | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- hrCTR Then No hrCTR: The experimental admission (hrCTR) was defined as having the participant complete a exercise session where the Diabetes Assistant (DiAs) Control-to-Range system is notified of heart rate. The study team member activated and deactivated a heart rate button when the subject's heart rate exceeded and then returned below 140 beats per minute.
  The admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
  heart rate Control to Range System (hrCTR) using DiAs Platform: Diabetes Assistant (DiAs) Medical Platform System
  * A smart-phone medical platform (DiAs);
  * Continuous Glucose Monitor;
  * Insulin pump;
  * Bluetooth connection;
  * Remote Monitoring Server.
  The control admission (no hrCTR) had participants complete an exercise session where the closed loop is not informed about heart rate.
  The admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
- No hrCTR Then hrCTR: The control admission (no hrCTR) had participants complete an exercise session where the closed loop is not informed about heart rate.
  The admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
  The experimental admission (hrCTR) was defined as having the participant complete a exercise session where the Diabetes Assistant (DiAs) Control-to-Range system is notified of heart rate. The study team member activated and deactivated a heart rate button when the subject's heart rate exceeded and then returned below 140 beats per minute.
  The admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
  heart rate Control to Range System (hrCTR) using DiAs Platform: Diabetes Assistant (DiAs) Medical Platform System
  * A smart-phone medical platform (DiAs);
  * Continuous Glucose Monitor;
  * Insulin pump;
  * Bluetooth connection;
  * Remote Monitoring Server.
- Total: Total of all reporting groups
Arm/Group | hrCTR Then No hrCTR | No hrCTR Then hrCTR | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [14 to 16] | 14 [13 to 16] | 14 [13 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
diabetes duration [y] [Median (Inter-Quartile Range); unit: years] | 10 [8 to 11.8] | 9 [6 to 13] | 10 [8 to 12.9]
HbA1c [%] [Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin] | 9.2 [8.3 to 9.7] | 8.7 [7.9 to 9.2] | 9.1 [8.2 to 9.6]
Total daily insulin [U] [Median (Inter-Quartile Range); unit: Units per day] | 62.5 [46 to 72] | 75 [50 to 80.2] | 65.1 [47.8 to 78.2]

OUTCOME MEASURES:

1. Primary Outcome: Low Blood Glucose Index (LBGI)
Description: The Low Blood Glucose Index, which quantifies the risk for hypoglycemia, and the hypoglycemic count (number sequences of blood glucose less than 70 mg/dL). The LBGI is a metric of the frequency and severity of hypoglycemia, based on an increasing weighting of progressively low glucose readings. The LBGI is measured on a scale from 0 to 100 and a higher score indicates a worse outcome.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: index score
Groups:
- hrCTR: The experimental admission (hrCTR) was defined as having the participant complete a exercise session where the Diabetes Assistant (DiAs) Control-to-Range system is notified of heart rate. The study team member activated and deactivated a heart rate button when the subject's heart rate exceeded and then returned below 140 beats per minute.
  The admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
- No hrCTR: The control admission (No hrCTR) had participants complete an exercise session where the closed loop is not informed about heart rate.
  The admission was about 24-hour in duration with at least 2 days of wash-out in between. Admission had to be completed within a 2-month window.
Arm/Group | hrCTR | No hrCTR
Number analyzed (Participants) | 18 | 18
index score | 1.4 (0.91) | 1.9 (1.85)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded once eligibility was met and was completed at the completion of the second admission (approximately 2 months).
Arm/Group | hrCTR | No hrCTR
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes